CLINICAL TRIAL: NCT07351955
Title: Clinical Study on a Novel Strategy of Individualized Non-Invasive Neuromodulation for the Treatment of Tic Disorders in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LY202504140
Record Dates: First submitted 2026-01-11; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Tic Disorders
Keywords: Transcranial Magnetic Stimulation
MeSH Terms: conditions — Tic Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The child will use a transcranial magnetic stimulator model ZL-N-010 to stimulate preselected targets located in the prefrontal lobe, bilateral temporal lobes, and parietal lobe. The child may rest as needed during the treatment process. Each TMS session lasts approximately 30 minutes. A total of 10 sessions will be administered. They will also use general behavioral therapy.
  Interventions: Device: Transcranial Magnetic Stimulation; Behavioral: general behavioral therapy
- Sham-Controlled Observation Group (Placebo Comparator): The child will receive sham stimulation and general behavioral therapy.
  Interventions: Behavioral: general behavioral therapy

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Transcranial magnetic stimulation (TMS) will be administered to the child using a ZL-N-010 model device, targeting predefined sites in the prefrontal, bilateral temporal, and parietal lobes.
  Arms: Intervention Group
Behavioral: general behavioral therapy — Behavioral interventions include avoiding screen time, parental avoidance of scolding or corporal punishment, and steering clear of activities or emotional stimuli that may exacerbate symptoms.

SUMMARY:
This study aims to establish a novel personalized closed-loop NiBS/TMS therapeutic strategy and clinical protocol for children with Tic Disorders (TDs) through a series of scientific investigations. Additionally, it seeks to elucidate the underlying neural circuit mechanisms, enhance the therapeutic efficacy of TMS in pediatric TDs, and achieve precision neuromodulation for children with TDs.

ELIGIBILITY:
Inclusion Criteria:

* 1: Children and adolescents aged 5 to 18 years

  2: Meets DSM-5 diagnostic criteria for Tic Disorders (TDs) with normal EEG findings

  3: No prior treatment received for TDs

  4: Full-scale intelligence quotient (FIQ) ≥70 on the Wechsler Intelligence Scale for Children-Revised (WISC-R)

Exclusion Criteria:

* 1: WISC-R Full-Scale Intelligence Quotient (FIQ) <70

  2: Presence of metal implants in the body ，Non-right-handedness

  3: Head movement (HM) >2mm during fMRI scanning, including both translational movement (TM) and rotational movement (RM)

  4: Any other neurological or psychiatric conditions, including but not limited to autism spectrum disorder (ASD), epilepsy, obsessive-compulsive disorder (OCD), etc

  5: Previous head trauma ，Neurological diseases ，Major systemic illnesses

Ages: 5 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Tic Severity | 10 weeks
  The severity of the child's clinical tic symptoms assessed via the Yale Global Tic Severity Scale.
Changes in brain region activation intensity and resting-state connectivity before and after treatment. | 10 weeks
  Based on fMRI imaging, changes in brain region activation intensity (BOLD signals) and resting-state functional connectivity (FC) before and after treatment were compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Children's Medical Center，School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No